CLINICAL TRIAL: NCT04308278
Title: Randomized, Placebo-controlled, Double Blind Study to Evaluate the Efficacy of 2LEBV® and 2LXFS® on Asthenia in Patients With an Epstein-Barr Virus Infection.
Brief Title: Study to Evaluate the Efficacy of 2LEBV® and 2LXFS® on Asthenia in Patients With an Epstein-Barr Virus Infection
Acronym: EBVAST
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Labo'Life (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LLB-2019-03
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2023-10

CONDITIONS: EBV Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2LEBV® / 2LXFS® (Experimental): 6 months of treatment
  Interventions: Drug: 2LEBV® / 2LXFS®
- Placebo (Placebo Comparator): 6 months of treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 2LEBV® / 2LXFS® — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: 2LEBV® / 2LXFS®
Drug: Placebo — The treatment schema consists in taking the content of one capsule a day, 15-30 minutes before breakfast, on an empty stomach, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment. The duration of treatment will be 6 months of continuous intake of the content of 1 capsule/day.
  Arms: Placebo

SUMMARY:
Worldwide, 95% of adults are infected with Epstein-Barr Virus (EBV). These infections may cause different diseases. In most cases, EBV infection is asymptomatic because of a highly effective host immune response. Some individuals develop infectious mononucleosis (a self-limiting lymphoproliferative disorder in adolescents and young adults that is considered to be the primary infection), while others develop chronic fatigue syndrome, EBV-associated lymphoid, or epithelial malignancies.

Today, there is no available treatment to treat and destroy EBV. The treatment is essentially symptomatic (treatment of the symptoms and not of the virus itself) with analgesics for pain for example.

The studied drugs are 2LEBV® and 2LXFS®, from Labo'Life company, and the treatment schema is the same for the two drugs: it consists in taking the content of one capsule per day, sequentially, according to capsules' numerical order: 1 through 10. When capsule number 10 is taken, capsule 1 of the next blister should be taken on the next day to continue the treatment.

The duration of treatment will be of 6 months of continuous intake of the content of 1 capsule/day.

The aim of this study is to provide additional information on effectiveness on the 2LEBV® and 2LXFS®in the treatment of EBV chronic and acute infections, and in particular to demonstrate their effectiveness versus placebo in the reduction of asthenia and other symptoms in EBV infection.

ELIGIBILITY:
Pré-Inclusion Criteria:

* Patients, male or female, aged 12 years and older,
* Patient with fatigue for 1 month or more,
* Patient with at least two other symptoms among the following: Long-lasting exhaustion even after light exertion, subfebrile state, fever, loss of appetite, nausea, angina, conjunctivis, sensitive cervical or axillary lymph nodes, erythematous and swollen tonsil, headaches, sore throat, myalgia, muscular weakness, arthralgia, splenomegaly, visual disorders, memory disorders, attention deficit disorders, sleep disorders, gastrointestinal disorders, breathing disorders, cardiovascular disorders.
* Patient (and/or parents if necessary) agrees to perform serology for the study,
* Patient (and/or parents if necessary) agrees to perform lymphocyte typing for the study during the pre-inclusion visit,
* Patients (and/or parents if necessary) having the faculties to understand and respect the constraints of the study,
* Signature of the Informed Consent Form by the patient (and/or parents if necessary).

Inclusion Criteria:

- Patient who have a positive serology for EBV (IgG and/or IgM positive).

Exclusion Criteria:

* Patient who have received any treatment with the 2LEBV® or 2LXFS®,
* Patients who have received any homeopathic treatment in the previous 2 months prior to the study,
* Patients under immunosuppressive treatment,
* Patient undergoing treatment for psychiatric disorders,
* Patients having received immunotherapy or micro-immunotherapy during the last 3 months,
* Patients with known lactose intolerance,
* Pregnant or breastfeeding women,
* Patients who participated in a clinical study in the previous 2-months period,
* Patients (and/or parents of patients if necessary) who are not sufficiently motivated to engage on the total study follow-up period, or likely to travel or to move before the end of the study,
* Patients with severe immunodeficiency disease requiring long term treatment (*) or patients under chemotherapy or radiotherapy,
* Patients under homeopathic or phytotherapy treatment,
* Patients addicted to or using recreational drugs,
* Patient under guardianship and/or curatorship, (*) important renal or respiratory insufficiency, transplanted or grafted patients, HIV/AIDS, terminal cancer.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Measure of the general fatigue scale of the Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire at the end of the treatment. | 6 months
  Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire. 5 scales. Higher scores means worse outcome.
  General Fatigue dimension: Minimum value: 4. Maximum Value: 20. Physical fatigue dimension: Minimum value: 4. Maximum Value: 20. Reduced activity dimension: Minimum value: 4. Maximum Value: 20. Reduced motivation dimension: Minimum value: 4. Maximum Value: 20. Mental fatigue dimension: Minimum value: 4. Maximum Value: 20.

SECONDARY OUTCOMES:
Comparison of the efficacy of the treatment on physical fatigue, reduced activity, reduced motivation and mental fatigue scales on the MFI-20 questionnaire between the 2LEBV® or the 2LXFS®/2LEBV® group versus the placebo group | 6 months
  Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire. 5 scales. Higher scores means worse outcome.
  Physical fatigue dimension: Minimum value: 4. Maximum Value: 20. Reduced activity dimension: Minimum value: 4. Maximum Value: 20. Reduced motivation dimension: Minimum value: 4. Maximum Value: 20. Mental fatigue dimension: Minimum value: 4. Maximum Value: 20.
Comparison of the efficacy of the treatment on general fatigue and other dimensions of the MFI-20 questionnaire between the 2LEBV® and the 2LXFS®/2LEBV® group versus the placebo group. | 3 months
  Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire. 5 scales. Higher scores means worse outcome.
  General Fatigue dimension: Minimum value: 4. Maximum Value: 20. Physical fatigue dimension: Minimum value: 4. Maximum Value: 20. Reduced activity dimension: Minimum value: 4. Maximum Value: 20. Reduced motivation dimension: Minimum value: 4. Maximum Value: 20. Mental fatigue dimension: Minimum value: 4. Maximum Value: 20.
Comparison of the efficacy of the treatment on general fatigue and other dimensions of the MFI-20 questionnaire between the 2LEBV® and the 2LXFS®/2LEBV® group versus the placebo group. | 12 months
  Multidiensional Fatigue Inventory-20 (MFI-20) questionnaire. 5 scales. Higher scores means worse outcome.
  General Fatigue dimension: Minimum value: 4. Maximum Value: 20. Physical fatigue dimension: Minimum value: 4. Maximum Value: 20. Reduced activity dimension: Minimum value: 4. Maximum Value: 20. Reduced motivation dimension: Minimum value: 4. Maximum Value: 20. Mental fatigue dimension: Minimum value: 4. Maximum Value: 20.
Comparisons of the efficacy of the treatment on others symptoms related to EBV infection and their duration between the 2LEBV® and 2LXFS®/2LEBV® group versus the placebo group. | 6 months
Comparisons of the efficacy of the treatment on others symptoms related to EBV infection and their duration between the 2LEBV® and 2LXFS®/2LEBV® group versus the placebo group. | 12 months
Comparison of the evolution of the lymphocytes typing between the 2LEBV® and 2LXFS®/2LEBV® group versus the placebo group. | 12 months
Safety: occurence of adverse events (AEs) and severe adverse events (SAEs), considered as related or not to the study drug. | 6 months
Comparisons of the efficacy of the treatment on others symptoms related to EBV infection and their duration between the 2LEBV® and 2LXFS®/2LEBV® group versus the placebo group. | 3 months

CONTACTS AND LOCATIONS:
Locations (11):
- Belgium (11):
  - Private Practice, Aartselaar
  - Private Practice, Boortmeerbeek
  - Private Practice, Brussels
  - Private practice, Brussels
  - Private Practice, Ghent
  - Private Practice, Jette
  - Private Practice, Limal
  - Private practice, Marche-en-Famenne
  - Cabinet privé, Schoten
  - Private practice, Stavelot
  - Private practice, Waregem

IPD SHARING:
Plan to Share IPD: No